CLINICAL TRIAL: NCT05557331
Title: Effectiveness of a Mobile App (PIMPmyHospital) in Reducing Therapeutic Turnaround Times in an Emergency Department: Protocol for a Pre-Post Intervention Study
Brief Title: Effectiveness of a Mobile App in Reducing Therapeutic TAT in an Emergency Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Clinical Research Platform (Other)
Responsible Party: Principal Investigator, Johan Siebert, MD, MD, Deputy Head of the Pediatric Emergency Department, Pediatric Emergency Physician, Pediatric Clinical Research Platform
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: PIMPmyHospital pre-post study
Record Dates: First submitted 2022-09-18; First posted 2022-09-28 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Emergency Medicine; Therapeutic Turnaround Time
Keywords: Information technologies; Mobile Applications; Laboratory Result Delivery; Therapeutic turnaround time; Information Storage and Retrieval; Hospital Communication Systems; Pediatric Emergency Medicine; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: A single center, non-equivalent comparison group, pre-post study.
Who Masked: Outcomes Assessor
Masking Description: Although neither the participants nor the study investigators can be blinded to the intervention, both will be blinded to the results of the study until their final analysis by the statistician. Participants will be informed only of the overall purpose of the study, which is to evaluate the effects of the app on quality of care, but not about the aim of reducing the time to access laboratory results to minimize bias. The statistician will remain blinded to allocation until the final analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-intervention (no app) (No Intervention): Participants before (12-month retrospective period) the implementation of the app in the emergency department.
- Post-intervention (PIMPmyHospital app) (Active Comparator): Participants that will use the mobile heath PIMPmyHospital app during the prospective 6-month period after the implementation of the app in the emergency department.
  Interventions: Device: PIMPmyHospital (mobile app)

INTERVENTIONS:
Device: PIMPmyHospital (mobile app) — After the implementation of the app, data will be collected prospectively over a 6-month period of use. This will include the times (HH:MM:SS) when the results issued by the central laboratory are made available on caregivers' mobile app and access times (as well as concurrent or preferred access times on the conventional computerized workstations should this occur).
  Arms: Post-intervention (PIMPmyHospital app)

SUMMARY:
This study is a single center, non-equivalent comparison group, pre-post study in a tertiary pediatric emergency department in Switzerland. the study will compare the control and experimental groups on outcome measures before (12-month period) and after (6-month period) the intervention consisting of the implementation and use of the evidence-based mobile app-the ''Patients In My Pocket in my Hospital'' (PIMPmyHospital) app.

The primary outcome will be the mean elapsed time in minutes between the delivery of lab results and the emergency department caregivers accessing them before (i.e., on the institutional electronic medical records) and after the implementation of the app (i.e, directly on the app).

DETAILED DESCRIPTION:
The study objective is to evaluate whether the use of the PIMPmyHospital app alters emergency departments (ED) physicians and nurses' temporal efficiency to learn about laboratory results more quickly while actively working in an ED. Temporal efficiency will be assessed by measuring the time between the release of the laboratory results in the clinical information system and their acknowledgement by these clinicians. Information regarding the app has been published previously (doi.org/10.3390/jpm12030428).

The investigators will conduct an 18-month, single center, non-equivalent comparison group, pre-post study. The study will compare the control and experimental groups on outcome measures before (12-month period) and after (6-month period) the intervention consisting of the use of the app. The study will take place in the pediatric ED of a tertiary referral and major trauma hospital in Switzerland, with an annual volume of 35,000 visits.

Eligible participants will be postgraduate residents pursuing a <6-year residency in pediatrics, pediatric emergency medicine fellows, and registered nurses from the pediatric ED (aged > 18 years). Written informed consent will be obtained from each participant in the interventional group after full information disclosure prior to study participation.

Before the implementation of the app, electronic medical records (EMR)-based data from the past 12 months will be collected retrospectively. These data include the times (i.e., HH:MM:SS) that results issued by the central laboratory were available on the institutional's EMR, as well as the times at which these results were accessed by caregivers via conventional computerized workstations. (ii) After the implementation of the app, data will be collected prospectively over a 6-month period of use. This will include the times (HH:MM:SS) when the results issued by the central laboratory are made available on caregivers' mobile app and access times, as well as concurrent or preferred access times on the conventional computerized workstations should this occur. Individual acceptance of the app on the first day (a priori), at 1 week, and then on the last day of the intervention (6 months) will be evaluated through the Unified Theory of Acceptance, and Use of Technology (UTAUT). Usability of the app will be measured by the System Usability Scale (SUS).

The primary outcome will be the mean elapsed time in minutes between the delivery of the lab results and the caregiver accessing them, both before and after the implementation of the app.

ELIGIBILITY:
Inclusion Criteria:

* Any postgraduate residents pursuing a <6 years residency in pediatrics.
* Any pediatric emergency medicine fellows.
* To be registered nurses from the pediatric emergency department.
* Participation agreement.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to lab results review | 1 year (retrospective) and 6 months (prospective)
  The mean elapsed time in minutes between the delivery of the lab results and the caregiver accessing them, both before and after the implementation of the app.

SECONDARY OUTCOMES:
Unified Theory of Acceptance, and Use of Technology (UTAUT) | 6 months
  Acceptance of the app by participants on the first day (a priori) and then at 1 week and on the last day of the intervention will be evaluated through the Unified Theory of Acceptance, and Use of Technology (UTAUT) questionnaire.
  The UTAUT is a 8-construct, 31-item questionnaire. The items are measure along a 5-point Likert scale, which ranges from "strongly agree" (1) to "strongly disagree" (5).
System Usability Scale (SUS) | 6 months
  Usability of the app will be measured by the System Usability Scale (SUS).
  The SUS comprises a 10-item questionnaire with 5 response options for each item based on their level of agreement, ranging from 1 (strongly disagree) to 5 (strongly agree). For odd-numbered statements (the positively worded items), the score contribution is equal to the scale position minus 1. For even-numbered statements (the negatively worded items), the score contribution is equal to 5 minus the scale position. Each score contribution falls within the range of 0 to 4. The participants' scores for each item are then added up together and multiplied by 2.5 to convert the original scores of 0 to 40 to 0 to 100. The higher the score, the better the usability.
Emergency department length of stay | 1 year (retrospective) and 6 months (prospective)
  The emergency department length of stay per patient measured from the point when patients are triaged in the ED to when discharged from the ED, defined as patients leaving the ED whether admitted to the intensive care unit or ward, transferred to another hospital for admission, discharged home, or those who left without being seen.
Cognitive alerts | 1 year (retrospective) and 6 months (prospective)
  Whether specific alerts, such as a flashing icon or sound for reported pathological values of laboratory results on the mobile app have an impact on the results.
  This will be measured using a questionnaire that each participant using the app will answer on a 5-point Likert scale, ranging from "strongly agree" (1) to "strongly disagree" (5).

CONTACTS AND LOCATIONS:
Overall Officials: Johan N Siebert, MD, Study Director — Geneva Children's Hospital, Geneva University Hospitals, Geneva, Switzerland
Locations (1):
- Geneva Children's Hospital, Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be deidentified and the study investigators will house the data locally on REDCap hosted on secured servers at the Geneva University Hospitals. The datasets used or analyzed during the current trial will be available from the corresponding author upon reasonable request, recognizing that these data will only provide results for the current pre-post study and not for future trials that would follow. Only deidentified/anonymized data will be shared.
Supporting Information: Study Protocol
Time Frame: Available from 6 month to 5 years after trial publication.
Access Criteria: * Data will be made available from the corresponding author upon approval of a proposal and with a signed data access agreement.
  * Deidentified participant data will be made available to qualified external researchers whose proposed use of the data has been approved by their Institutional Review Board.
  * Data will be made available for a specified research purpose.
  * The request proposal must include a statistician.

REFERENCES:
- [Background] Ehrler F, Tuor C, Rey R, Siebert JN. A Mobile App to Improve Patient Management in Emergency Departments: Caregiver Needs Analysis, Design and Early Technology Acceptance Assessment. Stud Health Technol Inform. 2021 Oct 27;285:233-238. doi: 10.3233/SHTI210605. PMID 34734879
- [Background] Ehrler F, Tuor C, Trompier R, Berger A, Ramusi M, Rey R, Siebert JN. Effectiveness of a Mobile App in Reducing Therapeutic Turnaround Time and Facilitating Communication between Caregivers in a Pediatric Emergency Department: A Randomized Controlled Pilot Trial. J Pers Med. 2022 Mar 9;12(3):428. doi: 10.3390/jpm12030428. PMID 35330427
- [Derived] Ehrler F, Tuor C, Rey R, Trompier R, Berger A, Ramusi M, Courvoisier DS, Siebert JN. Effectiveness of a Mobile App (PIMPmyHospital) in Reducing Therapeutic Turnaround Times in an Emergency Department: Protocol for a Pre- and Posttest Study. JMIR Res Protoc. 2023 May 3;12:e43695. doi: 10.2196/43695. PMID 37133909